CLINICAL TRIAL: NCT03591666
Title: A Non-randomized Phase II Study of Anlotinib in Recurrent/Metastatic Head and Neck Adenocarcinomas
Brief Title: A Study of Anlotinib in Recurrent/Metastatic Head and Neck Adenocarcinomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018HNRT02
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Head and Neck Carcinoma; Adenocarcinoma; Recurrent Disease; Distantly Metastatic Malignant Neoplasm
Keywords: head and neck adenocarcinoma; Anlotinib
MeSH Terms: conditions — Adenocarcinoma; Recurrence | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Anlotinib QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib p.o. qd

SUMMARY:
This is a non-randomized, phase II, open label study of anlotinib hydrochloride capsules in recurrent/metastatic adenocarcinomas of head and neck. The primary purpose of this study is to evaluate the efficacy of anlotinib.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed head and neck adenocarcinoma.
2. Patients with recurrent or metastatic head and neck adenocarcinoma who are not candidates for curative surgery or radiotherapy.
3. Measurable disease per the RECIST criteria.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
5. Provision of written informed consent.
6. Childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (IUD, birth control pills, or barrier device) during and for 3 months after completion of trial therapy.

Exclusion Criteria:

1. Prior treatment with Anlotinib
2. With pleural effusion or ascites, cause respiratory syndrome
3. Accepted the vascular endothelial growth inhibitor class targeted drug treatment of patients
4. Plan to take systemic anti-tumor therapy within 4 weeks before grouping or during the medicine-taking period of this research, including Cytotoxic Therapy, 5.Signal Transduction Inhibitor, and Immunotherapy (or who use Mitomycin C within 6 weeks before taking the treatment with experimental drug); The patients who have already taken Extended Field Radiotherapy (EF-RT) within 4 weeks before grouping or Limited Field Radiotherapy with proposed assessment of nidus within 2 weeks before grouping

6.Symptoms of brain metastases cannot be controlled and treated within less than 2 months 7.severe and failed to controlled diseases 8.Occurred venous thromboembolic events within 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2018-07-15 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months

SECONDARY OUTCOMES:
Progress free survival (PFS) | up to 24 months
Disease Control Rate (DCR) | up to 24 months
Overall Survival (OS) | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Guopei Zhu, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai ninth people's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No